CLINICAL TRIAL: NCT06414824
Title: The Impact of the isCGM Use on the Hypoglycemic Episodes and Fear of Hypoglycemia in Patients With Newly Diagnosed Type 1 Diabetes
Brief Title: The isCGM Use and Hypoglycemic Episodes and Fear of Hypoglycemia in Newly Diagnosed Type 1 Diabetes
Acronym: PENELOPE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study ended early due to CGM reimbursement policy changes, after that most patients eligible for the study could have isCGM reimbursed.
Sponsor: Jagiellonian University (Other)
Collaborators: Diabetes Poland (Unknown)
Responsible Party: Principal Investigator, Jerzy Hohendorff, MD, PhD, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PENELOPE
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: ambulatory glucose profile; time in range; fear of hypoglycemia; continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FreeStyle Libre (Experimental): FreeStyle Libre for 4 weeks.
  All subjects will wear a masked sensor (FreeStyle Libre Pro) for 14 days prior to randomisation.
  Interventions: Device: Intermittently Scanned Continuous Glucose Monitoring
- SMBG (Active Comparator): Subjects randomised to the control group will monitor their blood glucose with standard blood glucose meters.
  A 14-day FreeStyle Libre Pro is included for these subjects from day 14 to day 28 to collect glycaemic data for comparison to the intervention group of the study.
  All subjects will wear a masked sensor (FreeStyle Libre Pro) for 14 days prior to randomisation.
  Interventions: Device: Standard Blood Glucose Monitoring

INTERVENTIONS:
Device: Intermittently Scanned Continuous Glucose Monitoring — FreeStyle Libre, 4 weeks
  Other Names: FreeStyle Libre
  Arms: FreeStyle Libre
Device: Standard Blood Glucose Monitoring — Standard blood glucose monitoring with glucose meters
  Arms: SMBG

SUMMARY:
The aim of this trial is to investigate the impact of FreeStyle Libre use compared to SMBG on hypoglycemia episodes and fear of hypoglycemia in adults aged 18-35 with newly diagnosed type 1 diabetes.

This trial is conducted in university centers in Poland (Bialystok, Krakow, Poznan, Zabrze).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed type 1 diabetes (diagnosed based on the WHO criteria) no later than 6 months after the diagnosis.
* Insulin therapy: multiple daily injections,
* In the investigator's opinion, the participant must be technically capable of using the FreeStyle Libre system

Exclusion Criteria:

* Current or past use of any continuous glucose monitoring system.
* Pump therapy.
* Known allergy to medical adhesives.
* Oral steroid therapy.
* Pregnancy or planning pregnancy within the study duration.
* Breast feeding.
* Dialysis treatment.
* Having a pacemaker.
* Unstable coronary heart disease.
* Cystic fibrosis.
* Cancer.
* Psychiatric disorders.
* Severe end-organ damage (kidney, liver, etc) or any uncontrolled disorder.
* Hospitalization for any reason other than the newly diagnosed type 1 diabetes 6 months prior to inclusion.
* Participating in another clinical trial that could affect glucose measurements or glucose management.
* In the investigator's opinion, if the participant is considered unsuitable for inclusion in the study for any other reason.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Hypoglycemia Fear Survey II | Baseline and day 28
  Change in HFS II score from baseline to day 28
TBR <70 mg/dL | Baseline and days 14 to 28
  Difference in time <70 mg/dL between intervention and control group assessed in days 14 to 28

SECONDARY OUTCOMES:
TIR | Baseline and days 14 to 28
  Difference in TIR 70-180 mg/dL between intervention and control group assessed in days 14 to 28
TBR <54 mg/dL | Baseline and days 14 to 28
  Difference in TBR <54 mg/dL between intervention and control group assessed in days 14 to 28
TAR >180 mg/dl | Baseline and days 14 to 28
  Difference in TAR >180 mg/dL between intervention and control group assessed in days 14 to 28
TAR >250 mg/dl | Baseline and days 14 to 28
  Difference in TAR >250 mg/dL between intervention and control group assessed in days 14 to 28
DKA | Baseline to day 28
  Difference in number of hospitalizations for diabetic ketoacidosis between intervention and control group
Severe hypoglycemia | Baseline to day 28
  Difference in number of severe hypoglycemia episodes between intervention and control group
DDS | Baseline and day 28
  Change in DDS score from baseline to day 28
DTSQ | Baseline and day 28
  Change in DTSQ score from baseline to day 28
HFS II - Worry subscale | Baseline and day 28
  Change in HFS II - worry subscale from baseline to day 28
HFS II - Behaviour subscale | Baseline and day 28
  Change in HFS II - behaviour subscale from baseline to day 28

CONTACTS AND LOCATIONS:
Locations (4):
- Poland (4):
  - Department of Endocrinology, Diabetology and Internal Medicine, Medical University of Bialystok, Bialystok
  - Department of Metabolic Diseases, Jagiellonian University Medical College, Krakow
  - Department of Internal Medicine and Diabetology, Poznan University of Medical Sciences, Poznan
  - Department of Internal Medicine, Diabetology, and Cardiometabolic Disorders, Medical University of Silesia in Katowice, Zabrze

IPD SHARING:
Plan to Share IPD: No